CLINICAL TRIAL: NCT00491673
Title: A Prospective Randomized Trial of Uncemented Versus Cemented Hemiarthroplasty for Displaced Femoral Neck Fractures
Acronym: HEMI04
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Asker & Baerum Hospital (Other)
Responsible Party: Lars Nordsletten, Ulleval university hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEMI-SAB-UUS
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Femoral Neck Fractures
Keywords: Fracture; Femoral neck; Arthroplasty
MeSH Terms: conditions — Femoral Neck Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncemented (Active Comparator): Uncemented primary bipolar hemiarthroplasty of the hip
  Interventions: Procedure: Uncemented primary bipolar hemiarthroplasty of the hip
- Cemented (Active Comparator): Cemented primary bipolar hemiarthroplasty of the hip
  Interventions: Procedure: Cemented primary bipolar hemiarthroplasty of the hip

INTERVENTIONS:
Procedure: Uncemented primary bipolar hemiarthroplasty of the hip — Uncemented primary bipolar hemiarthroplasty of the hip
  Other Names: Corail, DePuy/Johnson and Johnson, United Kingdom
  Arms: Uncemented
Procedure: Cemented primary bipolar hemiarthroplasty of the hip — Cemented primary bipolar hemiarthroplasty of the hip
  Other Names: Spectron, Smith & Nephew, Memphis, TN
  Arms: Cemented

SUMMARY:
There is increasing evidence that primary hemiarthroplasty is the treatment of choice for displaced femoral neck fractures in the elderly

No definite conclusions have been made in regards to what kind of arthroplasty is favourable

Cemented implants are associated with increased risk of perioperative cardiovascular incidents and increased mortality.

Cementless implants are associated with increased postoperative pain and decreased walking ability.

This study investigates the differences between one well-documented cemented femoral stem and one well-documented uncemented femoral stem. Previous studies have mostly used uncemented stems with different designs.

Null hypothesis: No (less than 10 points) difference in HHS between groups at 1 year and 5 years

DETAILED DESCRIPTION:
Inclusion Criteria: Dislocated intracapsular femoral neck fracture in patients ≥ 70 years old Exclusion criteria: Pathological fracture, Systemic or local infection, Short life expectancy/not mobile at all, Symptomatic coxarthrosis.

Null hypothesis: No (less than 10 points) difference in HHS between groups at 1 year (SD of HHS is 15 points) Power: 95% Significance: 0.05 60 patients in each group needed. To compensate for high mortality and drop-out: 200 patients, 100 in each group

Randomized using www.randomization.org to create sealed opaque envelopes opened at inclusion after signed informed concent.

Recorded after surgery:

Operating time Arthroplasty components used Need of blood transfusion Blood loss Size of incision

Recorded at discharge, 3 months, 1 year and 5 years:

X-ray of pelvis and hip Harris Hip Score Barthels ADL-index Quality of life (EQ-5D) Use of analgetics Use of walking aids

Publication: International orthopaedic journal.

ELIGIBILITY:
Inclusion Criteria:

* Dislocated intracapsular femoral neck fracture
* ≥ 70 years old

Exclusion Criteria:

* Pathological fracture
* Systemic or local infection
* Short life expectancy/not mobile at all
* Symptomatic coxarthrosis

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2004-09; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome including pain (Harris Hip Score) | 5 years

SECONDARY OUTCOMES:
All Cause Mortality | 5 years
Activities Of Daily Living (Barthels ADL-Index) | 5 years
Quality Of Life (EQ-5D) | 5 years
Any treatment related complication | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Prof MD PhD, Study Chair — Ullevål University Hospital, University of Oslo; Wender Figved, MD, PhD, Principal Investigator — Asker and Baerum Hospital; Lars Nordsletten, Prof MD PhD, Study Director — Ullevål University Hospital, University of Oslo; Ellen Langslet, MD, Principal Investigator — Ullevaal University Hospital
Locations (2):
- Norway (2):
  - Ullevål University Hospital, Oslo, Oslo County
  - Sykehuset Asker And Baerum, Oslo, Rud

REFERENCES:
- See also: Pubmed link to publication of 1-year results — http://www.ncbi.nlm.nih.gov/pubmed/19130162